CLINICAL TRIAL: NCT03487822
Title: A Personalized Self-Management Program for Older Adults With Chronic Pain and Negative Emotions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1509016564; 28540451 (Other Grant/Funding Number: Pfizer)
Record Dates: First submitted 2018-03-19; First posted 2018-04-04 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Pain, Chronic; Negative Emotions
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The co-investigators performing assessments will be blind to the participant's arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Path Pain (Experimental): Path Pain participants will be receiving 8 weekly therapy session by license clinicians trained in the Path Pain intervention. Participants will also receive 4, 15-minute phone booster sessions, on a monthly basis after their final therapy session. Participants will also be invited to monthly group educational sessions. Both intervention and usual care participants will be receiving a pain educational booklet.
  Interventions: Behavioral: Path Pain
- Usual Care with Education (No Intervention): Usual Care with Education (UCE) will receive a pain educational booklet. Following completion of 24 weeks in the study, participants will also be invited to attend the monthly group educational sessions.
- Provider Feedback (No Intervention): Providers of patients in the study will take part in a short interview on their impressions of the intervention.

INTERVENTIONS:
Behavioral: Path Pain — The intervention examines the effects of PATH-Pain on emotion regulation to improve self-management of pain and pain-related disability in older adults with chronic pain, negative emotions, and cognitive impairment. This intervention consists of 8 weekly therapy sessions by a licensed clinician trained in Path Pain, 4 monthly boosters upon completion of therapy, and optional monthly group educational sessions.
  Arms: Path Pain

SUMMARY:
This study examines the effects of PATH-Pain on emotion regulation to improve self-management of pain and pain-related disability in older adults with chronic pain, negative emotions, and cognitive impairment. Half the participants will receive the intervention, and half the participants will receive usual care with education. Intervention subjects are hypothesized to have significantly less pain-related disability versus usual care subjects after 24 weeks.

DETAILED DESCRIPTION:
This study examines the effects of PATH-Pain on emotion regulation to improve self-management of pain and pain-related disability in older adults with chronic pain, negative emotions, and cognitive impairment. The investigators propose that emotion regulation is the mechanism of change through which PATH-Pain improves pain and pain-related disability (outcomes). This pilot study will provide initial evidence of the: a) feasibility and acceptability of PATH-Pain; b) effects of PATH-Pain on emotion regulation (mechanism of change) and outcomes (pain and pain-related disability); and c) mediating effect of emotion regulation (mechanism of change) on outcomes (pain and pain-related disability). The investigators will randomize 120 older adults (60 years or older) with chronic non-cancer related pain and negative emotions to PATH-Pain vs. Usual Care with Education (UCE). PATH-Pain will be administered by licensed mental health clinicians. Research assessments will be conducted at the Wright Center at study entry (baseline), and at 5, 10 (end of treatment), and 24 weeks.

Additionally, 20 providers of patients will be interviewed for feedback regarding the intervention.

Edits were made in November 2024 to better align with the study protocol regarding timing and measures.

ELIGIBILITY:
Inclusion Criteria

Patient Participants:

* 60 and older
* chronic pain (pain on most days in past 2 months)
* negative emotions
* MoCA score 16 or higher

Provider Participants:

* providers 18 or over that took care of patient participant

Exclusion Criteria - Patient Participants:

* MoCA score <16
* cancer related pain
* can not provide capacity to consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2019-07-26 (Actual); Study Completion 2019-07-26 (Actual)

PRIMARY OUTCOMES:
Change in Current Pain Intensity on an 11 point scale | Baseline, 10 weeks
  Pain intensity is an 11 item scale with a range of 0-11 with a higher score indicating higher pain.
Change in Pain-related disability (RMDQ) | Baseline, 10 weeks
  Pain-related disability as measured by the Roland-Morris Disability Questionnaire (RMDQ). This measure has a range of 0-24, with a higher score indicating higher disability.

SECONDARY OUTCOMES:
Change in Emotion Regulation Mediation (ERQ) | Baseline, 10 and 24 weeks
  The Emotion Regulation Questionnaire (ERQ) has a range of 7-70 with a higher score indicating higher emotion regulation strategy.
Client Satisfaction Questionnaire (CSQ) | 24 weeks
  Investigators will use 3 of the 8 questions in the Client Satisfaction Questionnaire (CSQ) which has a range of 3-12; a higher score indicating higher satifaction
Change in Montgomery-Asberg Depression Rating Scale (MADRS) | Baseline, 10 and 24 weeks
  The Montgomery-Asberg Depression Rating Scale (MADRS) has a range of 0-60 with a higher score indicating higher depression

CONTACTS AND LOCATIONS:
Overall Officials: Cary Reid, MD, PhD, Principal Investigator — Weill Medical College of Cornell University; Dimitris Kiosses, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Center on Aging (formerly Wright Center on Aging), New York, New York, United States